CLINICAL TRIAL: NCT01568892
Title: A Phase III Randomized, Double-blind Study to Demonstrate the Antiviral Activity of Dolutegravir (DTG) 50 mg Twice Daily Versus Placebo Both Co-Administered With a Failing Antiretroviral Regimen Over Seven Days, Followed by an Open Label Phase With All Subjects Receiving DTG 50 mg Twice Daily Co-administered With an Optimised Background Regimen (OBR) in HIV-1 Infected, Integrase Inhibitor Therapy-Experienced and Resistant, Adults
Brief Title: Study Assessing Dolutegravir in HIV-1 Infected Subjects With Virus Resistant to Raltegravir and/or Elivitegravir
Acronym: VIKING-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116529
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
Keywords: ART-experienced; GSK1349572; Integrase inhibitor resistance; Dolutegravir
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DTG 50 mg BID (Experimental): Subjects will receive dolutegravir (DTG) 50 milligrams (mg) twice daily (BID) and the components of their current failing antiretroviral regimen, except raltegravir or elvitegravir, for 7 days during the Double-blind (DB) Phase. From Day 8, all subjects will continue to receive DTG 50 mg BID with an optimized background regimen in the Open-label Phase.
  Interventions: Drug: Dolutegravir 50 mg twice daily
- Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase (Experimental): Subjects will receive matching placebo BID and the components of their current failing antiretroviral regimen, except raltegravir or elvitegravir, for 7 days during the DB Phase. From Day 8, all subjects will continue to receive DTG 50 mg BID with an optimized background regimen in the Open-label Phase.
  Interventions: Drug: Dolutegravir 50 mg twice daily; Drug: Dolutegravir placebo twice daily

INTERVENTIONS:
Drug: Dolutegravir 50 mg twice daily — Active dolutegravir plus failing background regimen (Day 1 to Day 7). Open label dolutegravir plus optimized background regimen (from Day 8)
  Other Names: GSK1349572
Drug: Dolutegravir placebo twice daily — Dolutegravir placebo plus failing background regimen (Day 1 to Day 7)
  Other Names: GSK1349572 Placebo
  Arms: Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase

SUMMARY:
Study ING116529 is a multicenter, randomized, study with an initial 7 day placebo- controlled, functional monotherapy phase to quantify the antiviral activity attributable to dolutegravir (DTG) in HIV-1 infected, ART-experienced adults who are experiencing virological failure on an Integrase inhibitor containing regimen (current RAL or ELV failures), with evidence of genotypic resistance to RAL or ELV at study entry. Thirty subjects will be randomized (1:1) to receive either DTG 50mg BID (Arm A) or Placebo (Arm B) with the current failing regimen for 7 days (RAL or ELV should be discontinued prior to dosing with DTG). At Day 8, subjects from both arms will enter an open label phase and receive open label DTG 50mg BID with an optimized background regimen containing at least one fully active drug.

DETAILED DESCRIPTION:
Study ING116529 is a multicenter, randomized, study with an initial 7 day placebo-controlled, functional monotherapy phase to assess the antiviral activity and safety of a dolutegravir (DTG, GSK1349572) containing regimen in HIV-1 infected, ART-experienced adults with virological failure on an integrase inhibitor (INI) containing regimen.

Subjects must have evidence of genotypic resistance to raltegravir [RAL] or elvitegravir [ELV] at Screening and documented current or historical genotypic or phenotypic resistance to at least two other antiretroviral therapy drug classes.

The study is designed to provide an accurate measure of the intrinsic antiviral activity of DTG 50mg twice daily versus placebo both administered with the current failing regimen in a randomised double-blind phase to Day 8. This will be followed by an open label phase with all subjects receiving DTG 50mg twice daily with an optimized background regimen (containing at least one fully active drug) until subjects no longer derive clinical benefit or until DTG is locally available. Thirty subjects will be randomized (1:1) to receive either DTG 50mg BID (Arm A) or Placebo (Arm B) with the current failing regimen for 7 days (RAL or ELV should be discontinued prior to dosing at Day 1). At Day 8, subjects from both arms will enter an open label phase and receive open label DTG 50mg BID with an optimized background regimen containing at least one fully active drug The primary analysis will be conducted after the last subject enrolled has completed the randomised, double-blind phase at Day 8. Additional analyses may be performed prior to study closure when all ongoing subjects transition to locally available commercial DTG.

ELIGIBILITY:
Inclusion Criteria:

* Screening plasma HIV-1 RNA ≥1000 copies/mL
* ART-experienced, INI-experienced, DTG naïve
* Current virological failure on raltegravir (RAL) or elvitegravir (ELV) regimen
* The subject's HIV-1 shows genotypic resistance to RAL or ELV at Screening
* Subject has been on stable ART for at least one month prior to Screening and through Day 1(with exceptions for ETV, EFV and NVP that can be interrupted within 14 days of Day 1, see Exclusion Criterion)
* Documented resistance to at least one drug from each of two or more of any approved classes of ART other than integrase inhibitors
* Be able to receive at least one fully active drug as part of the OBR from Day 8
* Women capable of becoming pregnant must use appropriate contraception during the study (as defined by the protocol)
* Willing and able to understand and provide signed and dated written informed consent prior to Screening.

Exclusion Criteria:

* Women who are pregnant or breast feeding
* An active AIDS-defining condition at Screening (except cutaneous Kaposi's sarcoma not requiring systemic therapy or CD4+ <200c/mm3)
* Moderate to severe hepatic impairment as defined by Child-Pugh classification
* Anticipated need for HCV therapy during the first 24 weeks of the study
* Recent history (less than or equal to 3 months) of any upper or lower gastrointestinal bleed, with the exception of anal or rectal bleeding
* Allergy or intolerance to the study drugs or their components or drugs of their class
* Malignancy within the past 6 months
* Treatment with an HIV-1 therapeutic vaccine within 90 days of Screening
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents or any immunomodulator within 28 days of Screening
* Treatment with any agent, other than licensed ART, with documented in vitro/vivo activity against HIV-1 within 28 days of first dose of investigational product (with the exception of entecavir if required for Hep B treatment)
* Treatment with etravirine, efavirenz, or nevirapine within 14 days of Day 1(etravirine may be used if coadministered with lopinavir/ritonavir or darunavir/ritonavir)
* Treatment with tipranivir/ritonavir, fosamprenavir, or fosamprenavir/ritonavir within 28 days prior to Screening
* Exposure to an experimental drug or vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, which ever is longer, prior to the first dose of IP.
* Any acute or verified Grade 4 laboratory abnormality (with the exception of Grade 4 lipids) at Screening
* ALT> 5 times the upper limit of normal (ULN) at Screening
* ALT ≥ 3X ULN and bilirubin > 1.5 X ULN (with 35% direct bilirubin) at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04-18 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2013-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (24):
- United States (24):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Annandale, Virginia

REFERENCES:
- [Derived] Akil B, Blick G, Hagins DP, Ramgopal MN, Richmond GJ, Samuel RM, Givens N, Vavro C, Song IH, Wynne B, Ait-Khaled M; VIKING-4 study team. Dolutegravir versus placebo in subjects harbouring HIV-1 with integrase inhibitor resistance associated substitutions: 48-week results from VIKING-4, a randomized study. Antivir Ther. 2015;20(3):343-8. doi: 10.3851/IMP2878. Epub 2014 Oct 16. PMID 25321146

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) meeting eligibility criteria at screening entered a 7-day randomized, double-blind, placebo-controlled phase. At Day 8, all par. entered an open-label phase and continued to receive dolutegravir with an optimized background regimen. A total of 75 par. were screened; 45 par. were screen failures, and 30 par. were randomized.
Groups:
- DTG 50 mg BID: Participants received dolutegravir (DTG) 50 milligrams (mg) twice daily (BID) and the components of their current failing antiretroviral regimen, except raltegravir or elvitegravir, for 7 days during the Double-blind (DB) Phase. From Day 8, all participants continued to receive DTG 50 mg BID with an optimized background regimen in the Open-label Phase.
- Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase: Participants received matching placebo BID and the components of their current failing antiretroviral regimen, except raltegravir or elvitegravir, for 7 days during the DB Phase. From Day 8, all participants continued to receive DTG 50 mg BID with an optimized background regimen in the Open-label Phase.
Period: Double-blind Phase
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Open-label Phase
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Started | 13 (One participant completing the DB Phase withdrew on Day 8 and did not enter the Open-label Phase.) | 16
Completed | 7 | 13
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 4 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (11.56) | 48.6 (8.85) | 48.1 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 8 | 8 | 16
  American Indian or Alaska Native | 0 | 1 | 1
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 4 | 7 | 11
  Missing: None of the Available Races Applied | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) at Day 8
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1) and Day 8. Change from Baseline was calculated as the value at Day 8 minus the value at Baseline (Day 1). The analysis was performed using statistical modeling correcting for Baseline plasma HIV-1 RNA, Baseline Dolutegravir (DTG) fold change (FC), the overall susceptibility score (OSS) of the failing regimen, and the interaction between DTG FC and treatment. Means and differences were calculated using the average Baseline DTG FC of the entire Intent-to-Treat Exposed (ITT-E) Population. The last observation carried forward with discontinuation equals Baseline (LOCFDB) dataset was used for the analysis. For the LOCFDB dataset, missing values were carried forward from the previous, non-missing, available on-treatment assessment, except formissing values due to premature withdrawal or Day 8 missing values, which had the Baseline value imputed.
Time Frame: Baseline and Day 8
Population: ITT-E Population: all randomized participants who received at least one dose of study medication. One participant receiving DTG 50 mg BID was excluded from analysis because they had no Baseline DTG FC value.
Measure: Least Squares Mean (Standard Error); unit: Log 10 copies per milliliter (c/mL)
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 13 | 16
Log 10 copies per milliliter (c/mL) | -1.06 (0.168) | 0.10 (0.183)
Statistical Analysis 1: Comparison: DTG 50 mg BID vs Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -1.16, 95% CI 2-sided [-1.52 to -0.80] — The estimated value represents the adjusted mean difference between the two treatment arms

2. Secondary Outcome: Absolute Values in Plasma HIV-1 RNA Over Time
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1), Day 8, Day 28, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, and Week 84. NA indicates data was not available.
Time Frame: Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72, and 84
Population: ITT-E Population. The Observed Case dataset, in which only the data that are available at a particular time point are used, with no imputation for missing values, was used for analysis. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Log10 c/mL
  Baseline, n=14, 16 | 4.02 (0.940) | 4.42 (0.760)
  Day 8, n=14, 16 | 2.95 (0.790) | 4.39 (0.844)
  Day 28, n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28, n=13, 16 | 2.14 (0.772) | 2.30 (1.054)
  Week 8, n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8, n=11, 16 | 2.35 (0.851) | 2.10 (0.913)
  Week 12, n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12, n=12, 14 | 2.51 (1.048) | 2.27 (1.179)
  Week 16, n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16, n=12, 16 | 2.57 (1.093) | 2.18 (1.098)
  Week 24, n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24, n=11, 15 | 2.65 (1.219) | 1.88 (0.654)
  Week 32, n=11, 14: number analyzed (Participants) | 11 | 14
  Week 32, n=11, 14 | 2.72 (1.176) | 1.81 (0.664)
  Week 40, n=7, 12: number analyzed (Participants) | 7 | 12
  Week 40, n=7, 12 | 2.35 (1.169) | 1.68 (0.133)
  Week 48, n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48, n=8, 13 | 2.47 (1.037) | 1.62 (0.088)
  Week 60, n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60, n=5, 12 | 2.15 (1.013) | 1.67 (0.150)
  Week 72, n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72, n=3, 4 | 2.35 (1.312) | 1.62 (0.054)
  Week 84, n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84, n=0, 1 |  | 1.59 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

3. Secondary Outcome: Mean Change From Baseline in Plasma HIV-1 RNA Over Time
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1), Day 8, Day 28, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, and Week 84. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72, and 84
Population: ITT-E Population. The Observed Case dataset, in which only the data that are available at the particular time point are used, with no imputation for missing values, was used for analysis. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Log10 c/mL
  Baseline, n=14, 16 | 4.02 (0.940) | 4.42 (0.760)
  Day 8, n=14, 16 | -1.07 (0.683) | -0.03 (0.262)
  Day 28, n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28, n=13, 16 | -1.87 (0.898) | -2.12 (1.111)
  Week 8, n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8, n=11, 16 | -1.89 (0.890) | -2.32 (1.112)
  Week 12, n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12, n=12, 14 | -1.54 (1.022) | -2.02 (1.245)
  Week 16, n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16, n=12, 16 | -1.48 (1.101) | -2.24 (1.180)
  Week 24, n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24, n=11, 15 | -1.38 (1.151) | -2.53 (1.033)
  Week 32, n=11, 14: number analyzed (Participants) | 11 | 14
  Week 32, n=11, 14 | -1.31 (1.059) | -2.62 (0.931)
  Week 40, n=7, 12: number analyzed (Participants) | 7 | 12
  Week 40, n=7, 12 | -1.48 (1.445) | -2.70 (0.843)
  Week 48, n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48, n=8, 13 | -1.34 (1.235) | -2.77 (0.881)
  Week 60, n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60, n=5, 12 | -1.91 (1.400) | -2.71 (0.863)
  Week 72, n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72, n=3, 4 | -2.08 (1.311) | -3.31 (0.968)
  Week 84, n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84, n=0, 1 |  | -3.75 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

4. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 c/mL Over Time
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1); Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, and 48. Number of participants with plasma HIV-1 RNA level <50 c/mL was obtained using Food and Drug Administration's (FDA's) snapshot algorithm, where all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) were treated as non-responders. Also, participants who switched their concomitant antiretroviral therapy (ART) prior to the visit of interest as follows were also treated as non-responders: background ART substitutions not permitted per protocol; background ART substitutions permitted per protocol; however, the decision to switch is not documented as being before or at the first On-treatment visit after switching to optimized background regimen (OBR) (i.e. Day 28) where HIV-1 RNA is assessed.
Time Frame: Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40 and 48
Population: ITT-E Population. The Snapshot dataset was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants
  Baseline | 0 | 0
  Day 8 | 1 | 0
  Day 28 | 6 | 6
  Week 8 | 5 | 9
  Week 12 | 6 | 8
  Week 16 | 5 | 8
  Week 24 | 6 | 8
  Week 32 | 4 | 9
  Week 40 | 4 | 7
  Week 48 | 3 | 9

5. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <400 c/mL Over Time
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1); Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40 and 48. Number of participants with plasma HIV-1 RNA level <400 c/mL was obtained using FDA's snapshot algorithm, where all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) were treated as non-responders. Also, participants who switch their concomitant ART prior to the visit of interest as follows were also treated as non-responders: background ART substitutions not permitted per protocol; background ART substitutions permitted per protocol; however the decision to switch is not documented as being before or at the first On-treatment visit after switching to OBR (i.e. Day 28) where HIV-1 RNA is assessed.
Time Frame: Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40 and 48
Population: ITT-E Population. The Snapshot dataset was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants
  Baseline | 2 | 0
  Day 8 | 4 | 0
  Day 28 | 9 | 12
  Week 8 | 7 | 13
  Week 12 | 7 | 10
  Week 16 | 7 | 12
  Week 24 | 6 | 11
  Week 32 | 6 | 10
  Week 40 | 5 | 10
  Week 48 | 6 | 10

6. Secondary Outcome: Absolute Values in Cluster of Differentiation 4+ (CD4+) Cell Counts Over Time
Description: Blood samples were collected for lymphocyte subset assessment by flow cytometry at Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72, and 84.
Time Frame: Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72, and 84
Population: ITT-E Population. The Observed Case dataset, in which only the data that are available at a particular time point are used, with no imputation for missing values, was used for analysis. Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeters
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Cells per cubic millimeters
  Baseline, n=14, 16 | 163.5 [111.0 to 231.0] | 90.5 [46.0 to 267.5]
  Day 8, n=14, 15: number analyzed (Participants) | 14 | 15
  Day 8, n=14, 15 | 198.5 [154.0 to 239.0] | 102.0 [50.0 to 310.0]
  Day 28, n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28, n=13, 16 | 174.0 [168.0 to 335.0] | 234.0 [114.5 to 303.5]
  Week 8, n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8, n=11, 16 | 211.0 [71.0 to 401.0] | 228.0 [124.0 to 357.5]
  Week 12, n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12, n=12, 14 | 223.5 [115.0 to 345.5] | 217.5 [121.0 to 333.0]
  Week 16, n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16, n=12, 16 | 241.0 [107.5 to 382.5] | 262.5 [132.5 to 436.5]
  Week 24, n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24, n=11, 15 | 232.0 [116.0 to 509.0] | 242.0 [194.0 to 399.0]
  Week 32, n=11, 14: number analyzed (Participants) | 11 | 14
  Week 32, n=11, 14 | 213.0 [91.0 to 489.0] | 326.0 [229.0 to 542.0]
  Week 40, n=8, 12: number analyzed (Participants) | 8 | 12
  Week 40, n=8, 12 | 299.5 [212.5 to 566.5] | 328.0 [204.5 to 508.0]
  Week 48, n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48, n=8, 13 | 328.0 [263.0 to 526.5] | 370.0 [231.0 to 457.0]
  Week 60, n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60, n=5, 12 | 321.0 [234.0 to 328.0] | 333.0 [217.5 to 541.0]
  Week 72, n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72, n=3, 4 | 321.0 [261.0 to 465.0] | 299.5 [231.5 to 349.0]
  Week 84, n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84, n=0, 1 |  | 368.0 [368.0 to 368.0]

7. Secondary Outcome: Median Change From Baseline in CD4+ Cell Counts Over Time
Description: Blood samples were collected for lymphocyte subset assessment by flow cytometry at Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72, and 84. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline; Day 8; Day 28; Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72, and 84
Population: ITT-E Population. Observed dataset was used for analysis. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeters
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Cells per cubic millimeters
  Baseline, n=14, 16 | 163.5 [111.0 to 231.0] | 90.5 [46.0 to 267.5]
  Day 8, n=14, 15: number analyzed (Participants) | 14 | 15
  Day 8, n=14, 15 | 7.0 [0.0 to 94.0] | 0.0 [-12.0 to 24.0]
  Day 28, n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28, n=13, 16 | 14.0 [6.0 to 68.0] | 68.5 [5.0 to 140.5]
  Week 8, n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8, n=11, 16 | 34.0 [10.0 to 96.0] | 87.5 [9.5 to 138.5]
  Week 12, n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12, n=12, 14 | 49.0 [-5.0 to 83.0] | 79.0 [1.0 to 121.0]
  Week 16, n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16, n=12, 16 | 76.5 [3.0 to 151.0] | 70.0 [20.5 to 235.0]
  Week 24, n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24, n=11, 15 | 39.0 [0.0 to 134.0] | 117.0 [23.0 to 163.0]
  Week 32, n=11, 14: number analyzed (Participants) | 11 | 14
  Week 32, n=11, 14 | 48.0 [0.0 to 198.0] | 135.5 [58.0 to 271.0]
  Week 40, n=8, 12: number analyzed (Participants) | 8 | 12
  Week 40, n=8, 12 | 90.5 [45.0 to 226.5] | 125.5 [50.0 to 244.5]
  Week 48, n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48, n=8, 13 | 115.0 [96.0 to 226.5] | 156.0 [68.0 to 293.0]
  Week 60, n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60, n=5, 12 | 170.0 [65.0 to 210.0] | 146.0 [73.5 to 242.0]
  Week 72, n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72, n=3, 4 | 163.0 [96.0 to 354.0] | 174.0 [147.0 to 225.0]
  Week 84, n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84, n=0, 1 |  | 269.0 [269.0 to 269.0]

8. Secondary Outcome: Absolute Values in Cluster of Differentiation 8+ (CD8+) Cell Counts Over Time
Description: Blood samples were collected for lymphocyte subset assessment by flow cytometry at Baseline; Day 28; and Weeks 12, 24, and 48.
Time Frame: Baseline; Day 28; Weeks 12, 24, and 48
Population: ITT-E Population. The Observed Case dataset, in which only the data that are available at a particular time point are used, with no imputation for missing values, was used for analysis. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Cells per cubic millimeter
  Baseline, n=14, 16 | 896.0 [589.0 to 1689.0] | 808.5 [436.5 to 1221.0]
  Day 28, n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28, n=13, 16 | 1135.0 [598.0 to 1741.0] | 973.0 [675.0 to 1322.0]
  Week 12, n=11, 14: number analyzed (Participants) | 11 | 14
  Week 12, n=11, 14 | 1198.0 [591.0 to 1977.0] | 1184.0 [860.0 to 1711.0]
  Week 24, n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24, n=11, 15 | 1160.0 [526.0 to 1908.0] | 1323.0 [969.0 to 1622.0]
  Week 48, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 48, n=6, 12 | 1295.0 [837.0 to 1818.0] | 1147.0 [753.0 to 1570.0]

9. Secondary Outcome: Median Change From Baseline in CD8+ Cell Counts Over Time
Description: Blood samples were collected for lymphocyte subset assessment by flow cytometry at Baseline; Day 28; and Weeks 12, 24, and 48. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline; Day 28; Weeks 12, 24, and 48
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Cells per cubic millimeter
  Baseline, n=14, 16 | 896.0 [589.0 to 1689.0] | 808.5 [436.5 to 1221.0]
  Day 28, n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28, n=13, 16 | 227.0 [-135.0 to 301.0] | 177.0 [51.0 to 278.5]
  Week 12, n=11, 14: number analyzed (Participants) | 11 | 14
  Week 12, n=11, 14 | 151.0 [-150.0 to 379.0] | 288.0 [193.0 to 484.0]
  Week 24, n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24, n=11, 15 | 79.0 [-183.0 to 269.0] | 543.0 [35.0 to 930.0]
  Week 48, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 48, n=6, 12 | 88.0 [-19.0 to 179.0] | 124.0 [-102.5 to 238.5]

10. Secondary Outcome: Number of Participants With the Indicated Type of HIV-1 Disease Progression (Acquired Immunodeficiency Syndrome [AIDS] or Death [DT])
Description: The number of participants with HIV-1 disease progression (AIDS or death) was assessed per the Centers for Disease Control and Prevention (CDC) 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. The CDC classifies HIV infection as Category A (participants with asymptomatic HIV infection, acute HIV infection with accompanying illness, or persistent generalized lymphadenopathy), Category B (participants with symptomatic non-AIDS condition, i.e., conditions that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection), and Category C (includes AIDS indicator conditions as defined by diagnostic or presumptive measures).
Time Frame: From the day of the first dose of study drug until early withdrawal or the Week 48 analysis cut-off date (median of 55 study weeks)
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants
  From CDC Class A to CDC Class C | 0 | 0
  From CDC Class B to CDC Class C | 0 | 0
  From CDC Class C to new CDC Class C | 0 | 0
  From CDC Class A, B, or C to Death | 2 | 0

11. Secondary Outcome: Number of Participants With Any Adverse Event (Serious and Non-serious) of the Indicated Grade
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in other situations. Adverse events were graded for severity according to the Division of AIDS (DAIDS) toxicity scales as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (potentially life threatening).
Time Frame: From the first dose of study medication until early withdrawal or through the Week 48 analysis data cut-off date (median of 55 study weeks)
Population: Safety Population: all randomized participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants
  Grade 1 | 0 | 4
  Grade 2 | 7 | 6
  Grade 3 | 2 | 3
  Grade 4 | 2 | 1

12. Secondary Outcome: Number of Participants With the Maximum Post-Baseline-emergent Clinical Chemistry Toxicities of the Indicated Grade
Description: Participants with post-Baseline-emergent clinical chemistry toxicities were analyzed. Clinical chemistry toxicities were graded for severity according to the DAIDS toxicity scales as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (potentially life threatening).
Time Frame: as for outcome 11
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants
  Grade 1 | 5 | 4
  Grade 2 | 5 | 5
  Grade 3 | 0 | 4
  Grade 4 | 0 | 1

13. Secondary Outcome: Number of Participants With the Maximum Post-Baseline-emergent Hematology Toxicities of the Indicated Grade
Description: Participants with post-Baseline-emergent hematology toxicities were analyzed. Hematology toxicities were graded for severity according to the DAIDS toxicity scales as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (potentially life threatening).
Time Frame: as for outcome 11
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants
  Grade 1 | 2 | 3
  Grade 2 | 2 | 5
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0

14. Secondary Outcome: AUC(0-tau) of DTG
Description: The area under the time concentration curve over the dosing interval (AUC[0-tau]) of DTG was assessed by a population pharmacokinetic (PK) modeling approach using pooled DTG PK data from multiple studies. Blood samples for the determination of plasma DTG concentration were collected at the following time points: pre-dose and 1-3 hours post-dose on Day 8; pre-dose and within a post-dose window (1-3 hours or 4-12 hours) on Day 28 and Week 24. For Day 8 PK, only samples collected from participants randomized to the active DTG arm were analyzed.
Time Frame: Day 8, Day 28, and Week 24
Population: PK concentration Population comprised of all participants who received DTG, underwent PK sampling during the study, and provided evaluable DTG plasma concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hour per mL (µg*hr/mL)
Groups:
- Overall Study Arm: All the participants who received DTG 50 mg BID.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 29
µg*hour per mL (µg*hr/mL) | 37.9 (41.8)

15. Secondary Outcome: Cmax of DTG
Description: The maximal concentration (Cmax) of DTG was assessed by a population PK modeling approach using pooled DTG PK data from multiple studies. Blood samples for the determination of plasma DTG concentration were collected at the following time points: pre-dose and 1-3 hours post-dose on Day 8; pre-dose and within a post-dose window (1-3 hours or 4-12 hours) on Day 28 and Week 24. For Day 8 PK, only samples collected from participants randomized to the active DTG arm were analyzed.
Time Frame: Day 8, Day 28, and Week 24
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (µg/mL)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 29
Micrograms per milliliter (µg/mL) | 4.14 (32.6)

16. Secondary Outcome: Plasma DTG Pre-dose Concentration (C0) at Day 8, Day 28, and Week 24; and Average DTG C0 (C0 Avg) at Week 24
Description: Blood samples for the determination of plasma DTG pre-dose concentration were collected pre-dose on Day 8, Day 28, and Week 24. For Day 8 PK, only samples collected from participants randomized to the active DTG arm were analyzed. C0 Avg was calculated at Week 24 as the mean of the concentration at Day 8, Day 28, and Week 24.
Time Frame: Day 8, Day 28, and Week 24
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 13 | 16
µg/mL
  Day 8 C0, n=10, 0: number analyzed (Participants) | 10 | 0
  Day 8 C0, n=10, 0 | 3.043 (44) |
  Day 28 C0, n=11, 16: number analyzed (Participants) | 11 | 16
  Day 28 C0, n=11, 16 | 1.393 (189) | 2.154 (81)
  Week 24 C0, n=10, 14: number analyzed (Participants) | 10 | 14
  Week 24 C0, n=10, 14 | 1.864 (110) | 2.201 (145)
  C0_avg, n=13, 16 | 1.820 (188) | 2.307 (76)

17. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Integrase (IN) Mutations Detected at the Time of Defined Virologic Failure (PDVF), as a Measure of Genotypic Resistance
Description: For participants meeting one of the criteria for PDVF, plasma samples collected at the time point of virologic failure were tested to evaluate any potential genotypic and/or phenotypic evolution of resistance. PDVF was defined as (A) Virologic Non-response: a decrease in plasma HIV-1 RNA of <1 log10 copies/mL by Day 28, with subsequent confirmation, unless plasma HIV-1 RNA is <400 copies/mL; confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 or (B) Virologic Rebound: confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL; confirmed plasma HIV-1 RNA levels >1 log10 copies/mL above the nadir value, where nadir is >=400 copies/mL.Treatment-emergent IN mutations are those detected at the time of PDVF but not at Baseline.
Time Frame: as for outcome 11
Population: PDVF Genotypic/Phenotypic Population: all participants in the ITT-E population with protocol-defined virologic failure. Only participants with Baseline integrase mutations with PDVF who had paired Baseline and time of PDVF samples were considered for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 5 | 2
Participants
  Any integrase mutation | 4 | 1
  L74L/M | 1 | 0
  T97A | 2 | 1
  E138E/K | 1 | 0
  E138K | 1 | 0
  S147G | 1 | 0
  N155N/H | 1 | 0

18. Secondary Outcome: Number of Participants With the Indicated Fold Increase in Fold Change (FC) in the 50% Inhibitory Concentration Relative to Wild-type Virus for DTG (i.e. PDVF FC/Baseline FC Ratio) at the Time of PDVF, as a Measure of Phenotypic Resistance
Description: For participants meeting one of the criteria for PDVF, plasma samples collected at the time point of virologic failure were tested to evaluate any potential genotypic and/or phenotypic evolution of resistance. The FC in IC50 (50% inhibitory concentration) for DTG relative to wild-type virus was determined for virus isolated at Baseline and at the time of PDVF. The number of participants with the indicated change (ratio) in the two values at the time of PDVF is presented. PDVF was defined as (A) Virologic Non-response: a decrease in plasma HIV-1 RNA of <1 log10 copies/mL by Day 28, with subsequent confirmation, unless plasma HIV-1 RNA is <400 copies/mL; confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 or (B) Virologic Rebound: confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL; confirmed plasma HIV-1 RNA levels >1 log10 copies/mL above the nadir value, where nadir is >=400 copies/mL.
Time Frame: as for outcome 11
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 5 | 2
Participants
  4-<8 fold increase in DTG FC | 0 | 1
  >=8 fold increase in DTG FC | 4 | 0

19. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AEs
Description: The number of participants who permanently discontinued study treatment due to AEs is presented.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Participants | 2 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Twelve lead ECG was performed using an automated ECG machine. The number of participants with abnormal-clinically significant ECG findings at any time on-treatment is reported.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants with data available at the specified time point was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 12 | 15
Participants | 1 | 1

21. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs including SBP and DBP were measured at Baseline, Week 24 and Week 48. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline and Weeks 24 and 48
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
millimeters of mercury
  SBP; Baseline; n=14, 16 | 120.4 (15.60) | 113.4 (9.99)
  SBP; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  SBP; Week 24; n=11, 15 | 2.0 (12.28) | 2.8 (13.82)
  SBP; Week 48; n=6, 12: number analyzed (Participants) | 6 | 12
  SBP; Week 48; n=6, 12 | -0.7 (19.50) | 3.1 (12.57)
  DBP; Baseline; n=14, 16 | 78.9 (12.51) | 75.1 (8.46)
  DBP; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  DBP; Week 24; n=11, 15 | -0.5 (9.49) | -1.2 (10.35)
  DBP; Week 48; n=6, 12: number analyzed (Participants) | 6 | 12
  DBP; Week 48; n=6, 12 | -1.2 (13.92) | -3.2 (8.78)

22. Secondary Outcome: Change From Baseline in Heart Rate
Description: Vital signs including heart rate was measured at Baseline, Week 24 and Week 48. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline and Weeks 24 and 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
beats per minute
  Baseline; n=14, 16 | 72.5 (9.70) | 75.9 (14.56)
  Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24; n=11, 15 | -1.4 (8.42) | 0.7 (11.20)
  Week 48; 6, 12: number analyzed (Participants) | 6 | 12
  Week 48; 6, 12 | 2.2 (11.03) | -2.5 (17.76)

23. Secondary Outcome: Change From Baseline in Albumin Level
Description: Blood samples were collected for the analysis of clinical chemistry parameters such as albumin. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline, Week 24 and 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
grams per liter
  Albumin; Baseline; n=14, 16 | 43.1 (4.13) | 43.4 (3.88)
  Albumin; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Albumin; Week 24; n=11, 15 | 0.0 (3.66) | 0.0 (3.87)
  Albumin; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Albumin; Week 48; n=8, 13 | 1.3 (2.55) | -0.8 (3.69)

24. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Creatine Kinase
Description: Blood samples were collected for the analysis of clinical chemistry parameters such as ALP, ALT, AST and creatine kinase. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
International units per liter
  ALP; Baseline; n=14, 16 | 91.9 (29.64) | 114.9 (106.74)
  ALP; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  ALP; Day 8; n=13, 15 | 1.9 (14.01) | -1.2 (9.41)
  ALP; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  ALP; Day 28; n=13, 16 | -6.1 (10.71) | -0.6 (11.37)
  ALP; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  ALP; Week 8; n=11, 16 | 1.6 (15.6) | 20.6 (63.97)
  ALP; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  ALP; Week 12; n=12, 14 | -0.8 (10.19) | -0.3 (26.15)
  ALP; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  ALP; Week 16; n=10, 16 | 3.1 (12.02) | 8.2 (40.55)
  ALP; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  ALP; Week 24; n=11, 15 | 1.7 (21.72) | 3.3 (54.06)
  ALP; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  ALP; Week 32; n=11, 14 | 6.9 (19.74) | 20.5 (35.89)
  ALP; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  ALP; Week 40; n=8, 12 | 2.3 (20.26) | 7.8 (24.69)
  ALP; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  ALP; Week 48; n=8, 13 | 28.0 (67.54) | 13.8 (32.07)
  ALP; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  ALP; Week 60; n=5, 12 | 6.0 (23.86) | 12.8 (35.98)
  ALP; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  ALP; Week 72; n=3, 4 | -5.0 (19.29) | 15.3 (10.21)
  ALP; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  ALP; Week 84; n=0, 1 |  | 22.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  ALT; Baseline; n=14, 16 | 24.9 (13.33) | 37.4 (22.70)
  ALT; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  ALT; Day 8; n=13, 15 | 0.0 (7.02) | -3.8 (11.91)
  ALT; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  ALT; Day 28; n=13, 16 | 0.4 (15.45) | -5.3 (23.65)
  ALT; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  ALT; Week 8; n=11, 16 | 1.2 (20.30) | -9.2 (17.93)
  ALT; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  ALT; Week 12; n=12, 14 | -5.4 (4.94) | -8.7 (23.36)
  ALT; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  ALT; Week 16; n=10, 16 | -5.2 (3.97) | -10.1 (23.02)
  ALT; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  ALT; Week 24; n=11, 15 | 3.1 (18.66) | -14.5 (23.16)
  ALT; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  ALT; Week 32; n=11, 14 | 0.9 (14.01) | -10.6 (25.77)
  ALT; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  ALT; Week 40; n=8, 12 | -1.6 (8.75) | -7.7 (25.86)
  ALT; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  ALT; Week 48; n=8, 13 | 7.9 (20.02) | -9.2 (23.50)
  ALT; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  ALT; Week 60; n=5, 12 | 0.8 (7.19) | -8.3 (24.28)
  ALT; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  ALT; Week 72; n=3, 4 | 8.7 (17.67) | -29.3 (33.06)
  ALT; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  ALT; Week 84; n=0, 1 |  | -3.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  AST; Baseline; n=14, 16 | 28.9 (11.13) | 34.9 (14.35)
  AST; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  AST; Day 8; n=13, 15 | 1.0 (11.50) | -2.0 (9.17)
  AST; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  AST; Day 28; n=13, 16 | -4.0 (10.13) | -2.3 (17.08)
  AST; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  AST; Week 8; n=11, 16 | -2.9 (7.57) | -6.3 (9.64)
  AST; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  AST; Week 12; n=12, 14 | -4.8 (4.07) | -5.1 (11.78)
  AST; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  AST; Week 16; n=10, 16 | -4.0 (2.94) | -6.6 (12.27)
  AST; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  AST; Week 24; n=11, 15 | 1.7 (14.05) | -10.1 (11.87)
  AST; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  AST; Week 32; n=11, 14 | -1.7 (6.83) | -7.4 (13.14)
  AST; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  AST; Week 40; n=8, 12 | -4.9 (4.09) | -4.1 (12.46)
  AST; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  AST; Week 48; n=8, 13 | 9.0 (27.77) | -5.4 (10.47)
  AST; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  AST; Week 60; n=5, 12 | -3.2 (1.64) | -5.9 (9.24)
  AST; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  AST; Week 72; n=3, 4 | 1.3 (8.50) | -13.8 (12.31)
  AST; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  AST; Week 84; n=0, 1 |  | -8.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Creatine Kinase; Baseline; n=14, 16 | 162.4 (129.21) | 130.3 (76.46)
  Creatine Kinase; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Creatine Kinase; Day 8; n=13, 15 | -2.1 (122.28) | -1.5 (53.29)
  Creatine Kinase; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Creatine Kinase; Day 28; n=13, 16 | -35.6 (96.22) | 37.0 (123.10)
  Creatine Kinase; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Creatine Kinase; Week 8; n=11, 16 | -16.4 (106.99) | -7.3 (68.19)
  Creatine Kinase; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Creatine Kinase; Week 12; n=12, 14 | -18.8 (105.64) | 0.4 (84.85)
  Creatine Kinase; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Creatine Kinase; Week 16; n=10, 16 | 34.2 (81.44) | 80.5 (305.19)
  Creatine Kinase; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Creatine Kinase; Week 24; n=11, 15 | -24.4 (82.07) | -6.0 (67.29)
  Creatine Kinase; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Creatine Kinase; Week 32; n=11, 14 | 2.3 (54.41) | 23.4 (96.88)
  Creatine Kinase; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Creatine Kinase; Week 40; n=8, 12 | -50.0 (93.45) | 66.3 (168.54)
  Creatine Kinase; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Creatine Kinase; Week 48; n=8, 13 | 7.8 (71.57) | 16.1 (68.96)
  Creatine Kinase; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Creatine Kinase; Week 60; n=5, 12 | -12.2 (23.30) | 18.8 (86.19)
  Creatine Kinase; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Creatine Kinase; Week 72; n=3, 4 | 35.0 (68.61) | -29.0 (76.27)
  Creatine Kinase; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Creatine Kinase; Week 84; n=0, 1 |  | -134.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

25. Secondary Outcome: Change From Baseline in Total Bilirubin (T. Bil) and Creatinine Levels
Description: Blood samples were collected for the analysis of clinical chemistry parameters such as T. Bil and creatinine. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Micromoles per liter
  T. Bil.; Baseline; n=14, 16 | 10.0 (4.51) | 7.5 (3.14)
  T. Bil.; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  T. Bil.; Day 8; n=13, 15 | 0.8 (6.81) | -1.1 (2.12)
  T. Bil.; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  T. Bil.; Day 28; n=13, 16 | -0.2 (6.19) | 2.1 (9.78)
  T. Bil.; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  T. Bil.; Week 8; n=11, 16 | 0.0 (4.20) | 3.1 (13.76)
  T. Bil.; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  T. Bil.; Week 12; n=12, 14 | 0.5 (4.76) | -0.6 (2.14)
  T. Bil.; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  T. Bil.; Week 16; n=10, 16 | 0.6 (3.89) | 1.9 (10.89)
  T. Bil.; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  T. Bil.; Week 24; n=11, 15 | 0.2 (2.89) | 2.1 (8.19)
  T. Bil.; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  T. Bil.; Week 32; n=11, 14 | -0.4 (3.20) | 2.3 (10.16)
  T. Bil.; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  T. Bil.; Week 40; n=8, 12 | 0.0 (3.70) | 3.3 (12.43)
  T. Bil.; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  T. Bil.; Week 48; n=8, 13 | -0.8 (4.13) | 3.2 (12.18)
  T. Bil.; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  T. Bil.; Week 60; n=5, 12 | -2.4 (2.61) | 2.3 (11.63)
  T. Bil.; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  T. Bil.; Week 72; n=3, 4 | -1.3 (4.16) | 9.5 (16.36)
  T. Bil.; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  T. Bil.; Week 84; n=0, 1 |  | 2.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Creatinine; Baseline; n=14, 16 | 86.94 (18.971) | 88.96 (24.013)
  Creatinine; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Creatinine; Day 8; n=13, 15 | 10.96 (24.505) | 0.11 (14.873)
  Creatinine; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Creatinine; Day 28; n=13, 16 | 12.72 (19.697) | 13.58 (21.030)
  Creatinine; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Creatinine; Week 8; n=11, 16 | 12.15 (8.570) | 15.79 (19.574)
  Creatinine; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Creatinine; Week 12; n=12, 14 | 6.86 (9.153) | 9.85 (13.274)
  Creatinine; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Creatinine; Week 16; n=10, 16 | 8.22 (13.464) | 7.68 (13.031)
  Creatinine; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Creatinine; Week 24; n=11, 15 | 1.63 (11.098) | 13.31 (17.347)
  Creatinine; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Creatinine; Week 32; n=11, 14 | 0.98 (7.441) | 15.96 (11.902)
  Creatinine; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Creatinine; Week 40; n=8, 12 | 3.58 (10.788) | 12.94 (13.870)
  Creatinine; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Creatinine; Week 48; n=8, 13 | 4.21 (19.450) | 12.85 (9.128)
  Creatinine; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Creatinine; Week 60; n=5, 12 | 4.96 (5.560) | 11.72 (15.820)
  Creatinine; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Creatinine; Week 72; n=3, 4 | 0.93 (8.529) | 13.25 (16.957)
  Creatinine; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Creatinine; Week 84; n=0, 1 |  | 1.80 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

26. Secondary Outcome: Change From Baseline in Cholesterol, Chloride, Carbon Dioxide (CO2)/Bicarbonate (HCO3), Glucose, High Density Lipoprotein Cholesterol, Potassium, Low Density Lipoprotein (LDL) Cholesterol, Sodium, Phosphorus, Triglycerides and Urea/Blood Urea Nitrogen
Description: Blood samples were collected for the analysis of clinical chemistry parameters such as cholesterol, chloride, CO2/HCO3, glucose, high density lipoprotein (HDL) cholesterol, potassium, LDL cholesterol, sodium, phosphorus inorganic, triglycerides and urea/blood urea nitrogen (BUN). Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: Safety Population. Lipid and glucose parameters were only summarized on fasting data. Only those participants available at the specified time points were analyzed (represented by n=X in category titles)
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Millimoles per liter
  Cholesterol; Baseline; n=8, 10: number analyzed (Participants) | 8 | 10
  Cholesterol; Baseline; n=8, 10 | 3.819 (0.9219) | 4.725 (1.7430)
  Cholesterol; Week 12; n=6, 8: number analyzed (Participants) | 6 | 8
  Cholesterol; Week 12; n=6, 8 | 0.433 (0.4622) | 0.538 (0.9598)
  Cholesterol; Week 24; n=6, 10: number analyzed (Participants) | 6 | 10
  Cholesterol; Week 24; n=6, 10 | 0.308 (0.3137) | 0.585 (1.0296)
  Cholesterol; Week 48; n=3, 7: number analyzed (Participants) | 3 | 7
  Cholesterol; Week 48; n=3, 7 | 0.567 (0.2021) | 0.421 (1.2770)
  Cholesterol; Week 60; n=2, 5: number analyzed (Participants) | 2 | 5
  Cholesterol; Week 60; n=2, 5 | 0.375 (0.9546) | -0.020 (1.3326)
  Cholesterol; Week 72; n=0, 1: number analyzed (Participants) | 0 | 1
  Cholesterol; Week 72; n=0, 1 |  | 1.350 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Chloride; Baseline; n=14, 16 | 104.1 (1.59) | 105.4 (3.32)
  Chloride; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Chloride; Day 8; n=13, 15 | 0.5 (1.61) | 0.4 (2.03)
  Chloride; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Chloride; Day 28; n=13, 16 | 0.4 (2.26) | -0.5 (2.58)
  Chloride; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Chloride; Week 8; n=11, 16 | 0.5 (1.97) | -1.8 (3.08)
  Chloride; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Chloride; Week 12; n=12, 14 | -0.8 (1.71) | 0.1 (2.73)
  Chloride; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Chloride; Week 16; n=10, 16 | 1.4 (1.90) | -1.0 (2.73)
  Chloride; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Chloride; Week 24; n=11, 15 | 0.9 (1.45) | -1.2 (3.14)
  Chloride; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Chloride; Week 32; n=11, 14 | 1.1 (2.21) | 0.0 (2.57)
  Chloride; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Chloride; Week 40; n=8, 12 | 0.5 (2.51) | 1.3 (2.80)
  Chloride; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Chloride; Week 48; n=8, 13 | 1.5 (3.74) | -0.1 (3.38)
  Chloride; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Chloride; Week 60; n=5, 12 | 2.0 (2.12) | 1.1 (2.81)
  Chloride; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Chloride; Week 72; n=3, 4 | 2.0 (2.65) | 1.0 (2.94)
  Chloride; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Chloride; Week 84; n=0, 1 |  | -2.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  CO2/HCO3; Baseline; n=14, 16 | 22.5 (2.07) | 20.8 (4.12)
  CO2/HCO3; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  CO2/HCO3; Day 8; n=13, 15 | 0.2 (1.30) | 0.1 (2.25)
  CO2/HCO3; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  CO2/HCO3; Day 28; n=13, 16 | 0.4 (2.29) | 1.1 (2.47)
  CO2/HCO3; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  CO2/HCO3; Week 8; n=11, 16 | 1.2 (1.66) | 1.6 (3.40)
  CO2/HCO3; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  CO2/HCO3; Week 12; n=12, 14 | 1.7 (1.92) | 1.9 (2.73)
  CO2/HCO3; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  CO2/HCO3; Week 16; n=10, 16 | -0.2 (2.39) | 1.8 (3.42)
  CO2/HCO3; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  CO2/HCO3; Week 24; n=11, 15 | 0.9 (1.92) | 1.5 (2.92)
  CO2/HCO3; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  CO2/HCO3; Week 32; n=11, 14 | 1.5 (2.21) | 0.8 (2.69)
  CO2/HCO3; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  CO2/HCO3; Week 40; n=8, 12 | 0.9 (2.30) | -0.2 (2.25)
  CO2/HCO3; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  CO2/HCO3; Week 48; n=8, 13 | -0.4 (2.13) | 1.7 (3.01)
  CO2/HCO3; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  CO2/HCO3; Week 60; n=5, 12 | 0.8 (1.30) | 0.3 (2.42)
  CO2/HCO3; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  CO2/HCO3; Week 72; n=3, 4 | 2.0 (3.61) | -0.3 (1.89)
  CO2/HCO3; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  CO2/HCO3; Week 84; n=0, 1 |  | 4.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Glucose; Baseline; n=12, 16: number analyzed (Participants) | 12 | 16
  Glucose; Baseline; n=12, 16 | 4.84 (0.535) | 5.56 (1.994)
  Glucose; Week 12; n=11, 14: number analyzed (Participants) | 11 | 14
  Glucose; Week 12; n=11, 14 | -0.01 (0.677) | 0.04 (0.679)
  Glucose; Week 24; n=10, 15: number analyzed (Participants) | 10 | 15
  Glucose; Week 24; n=10, 15 | 0.17 (0.957) | -0.08 (1.024)
  Glucose; Week 48; n=7, 13: number analyzed (Participants) | 7 | 13
  Glucose; Week 48; n=7, 13 | 0.13 (0.439) | 0.40 (1.143)
  Glucose; Week 60; n=3, 12: number analyzed (Participants) | 3 | 12
  Glucose; Week 60; n=3, 12 | 0.20 (0.300) | -0.18 (0.723)
  Glucose; Week 72; n=2, 4: number analyzed (Participants) | 2 | 4
  Glucose; Week 72; n=2, 4 | 0.45 (0.071) | 0.20 (0.744)
  HDL Cholesterol; Baseline; n=8, 10: number analyzed (Participants) | 8 | 10
  HDL Cholesterol; Baseline; n=8, 10 | 0.956 (0.2718) | 1.090 (0.2846)
  HDL Cholesterol; Week 12; n=6, 8: number analyzed (Participants) | 6 | 8
  HDL Cholesterol; Week 12; n=6, 8 | 0.117 (0.0683) | 0.156 (0.2485)
  HDL Cholesterol; Week 24; n=6, 10: number analyzed (Participants) | 6 | 10
  HDL Cholesterol; Week 24; n=6, 10 | 0.025 (0.1864) | 0.130 (0.2573)
  HDL Cholesterol; Week 48; n=3, 7: number analyzed (Participants) | 3 | 7
  HDL Cholesterol; Week 48; n=3, 7 | 0.117 (0.1155) | 0.136 (0.3363)
  HDL Cholesterol; Week 60; n=2, 5: number analyzed (Participants) | 2 | 5
  HDL Cholesterol; Week 60; n=2, 5 | -0.025 (0.0354) | 0.010 (0.3896)
  HDL Cholesterol; Week 72; n=0, 1: number analyzed (Participants) | 0 | 1
  HDL Cholesterol; Week 72; n=0, 1 |  | 0.350 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Potassium; Baseline; n=14, 16 | 4.16 (0.420) | 4.13 (0.377)
  Potassium; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Potassium; Day 8; n=13, 15 | -0.09 (0.198) | -0.01 (0.301)
  Potassium; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Potassium; Day 28; n=13, 16 | 0.19 (0.439) | 0.14 (0.518)
  Potassium; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Potassium; Week 8; n=11, 16 | 0.12 (0.379) | 0.19 (0.421)
  Potassium; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Potassium; Week 12; n=12, 14 | 0.03 (0.253) | 0.06 (0.373)
  Potassium; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Potassium; Week 16; n=10, 16 | -0.06 (0.360) | -0.08 (0.556)
  Potassium; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Potassium; Week 24; n=11, 15 | 0.17 (0.374) | 0.27 (0.641)
  Potassium; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Potassium; Week 32; n=11, 14 | -0.04 (0.329) | 0.27 (0.327)
  Potassium; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Potassium; Week 40; n=8, 12 | -0.01 (0.189) | 0.12 (0.259)
  Potassium; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Potassium; Week 48; n=8, 13 | 0.15 (0.532) | 0.28 (0.508)
  Potassium; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Potassium; Week 60; n=5, 12 | 0.06 (0.288) | 0.03 (0.614)
  Potassium; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Potassium; Week 72; n=3, 4 | 0.37 (0.208) | 0.02 (0.512)
  Potassium; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Potassium; Week 84; n=0, 1 |  | 0.20 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  LDL Cholesterol; Baseline; n=8, 9: number analyzed (Participants) | 8 | 9
  LDL Cholesterol; Baseline; n=8, 9 | 2.218 (0.9134) | 2.591 (1.3696)
  LDL Cholesterol; Week 12; n=6, 8: number analyzed (Participants) | 6 | 8
  LDL Cholesterol; Week 12; n=6, 8 | 0.293 (0.4197) | 0.500 (0.5145)
  LDL Cholesterol; Week 24; n=6, 9: number analyzed (Participants) | 6 | 9
  LDL Cholesterol; Week 24; n=6, 9 | 0.032 (0.5854) | 0.596 (0.7389)
  LDL Cholesterol; Week 48; n=3, 6: number analyzed (Participants) | 3 | 6
  LDL Cholesterol; Week 48; n=3, 6 | 0.330 (0.0458) | 0.322 (0.7725)
  LDL Cholesterol; Week 60; n=2, 4: number analyzed (Participants) | 2 | 4
  LDL Cholesterol; Week 60; n=2, 4 | 0.125 (0.5303) | -0.008 (1.0682)
  LDL Cholesterol; Week 72; n=0, 1: number analyzed (Participants) | 0 | 1
  LDL Cholesterol; Week 72; n=0, 1 |  | 1.110 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Sodium; Baseline; n=14, 16 | 138.8 (2.26) | 138.5 (2.22)
  Sodium; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Sodium; Day 8; n=13, 15 | 0.2 (1.64) | -0.1 (2.02)
  Sodium; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Sodium; Day 28; n=13, 16 | -0.2 (3.11) | -0.4 (2.60)
  Sodium; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Sodium; Week 8; n=11, 16 | 0.2 (2.14) | -0.4 (2.03)
  Sodium; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Sodium; Week 12; n=12, 14 | -0.5 (1.88) | 0.4 (2.53)
  Sodium; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Sodium; Week 16; n=10, 16 | 1.3 (2.06) | 0.2 (1.94)
  Sodium; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Sodium; Week 24; n=11, 15 | 0.5 (1.51) | -0.1 (2.33)
  Sodium; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Sodium; Week 32; n=11, 14 | 0.8 (1.60) | 0.1 (1.41)
  Sodium; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Sodium; Week 40; n=8, 12 | 1.0 (2.14) | 0.5 (1.57)
  Sodium; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Sodium; Week 48; n=8, 13 | 0.9 (3.56) | 0.9 (2.40)
  Sodium; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Sodium; Week 60; n=5, 12 | 2.4 (1.95) | 0.7 (2.46)
  Sodium; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Sodium; Week 72; n=3, 4 | 1.3 (2.52) | 0.3 (1.50)
  Sodium; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Sodium; Week 84; n=0, 1 |  | 0.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Phosphorus, inorganic; Baseline; n=14, 16 | 1.018 (0.1552) | 1.128 (0.1390)
  Phosphorus, inorganic; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Phosphorus, inorganic; Day 8; n=13, 15 | 0.012 (0.1261) | -0.123 (0.1635)
  Phosphorus, inorganic; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Phosphorus, inorganic; Day 28; n=13, 16 | 0.065 (0.2357) | -0.075 (0.1713)
  Phosphorus, inorganic; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Phosphorus, inorganic; Week 8; n=11, 16 | 0.018 (0.1722) | -0.075 (0.2244)
  Phosphorus, inorganic; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Phosphorus, inorganic; Week 12; n=12, 14 | 0.033 (0.1542) | -0.054 (0.1322)
  Phosphorus, inorganic; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Phosphorus, inorganic; Week 16; n=10, 16 | 0.080 (0.2263) | -0.053 (0.2617)
  Phosphorus, inorganic; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Phosphorus, inorganic; Week 24; n=11, 15 | -0.050 (0.1204) | -0.023 (0.1954)
  Phosphorus, inorganic; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Phosphorus, inorganic; Week 32; n=11, 14 | -0.036 (0.1343) | -0.050 (0.1787)
  Phosphorus, inorganic; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Phosphorus, inorganic; Week 40; n=8, 12 | 0.000 (0.1035) | -0.046 (0.2340)
  Phosphorus, inorganic; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Phosphorus, inorganic; Week 48; n=8, 13 | 0.025 (0.1282) | -0.031 (0.1331)
  Phosphorus, inorganic; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Phosphorus, inorganic; Week 60; n=5, 12 | 0.020 (0.1304) | -0.042 (0.1311)
  Phosphorus, inorganic; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Phosphorus, inorganic; Week 72; n=3, 4 | 0.017 (0.1258) | 0.013 (0.1031)
  Phosphorus, inorganic; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Phosphorus, inorganic; Week 84; n=0, 1 |  | 0.100 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Triglycerides; Baseline; n=8, 10: number analyzed (Participants) | 8 | 10
  Triglycerides; Baseline; n=8, 10 | 1.410 (0.5005) | 2.336 (1.1103)
  Triglycerides; Week 12; n=6, 8: number analyzed (Participants) | 6 | 8
  Triglycerides; Week 12; n=6, 8 | 0.047 (0.6380) | -0.260 (1.1159)
  Triglycerides; Week 24; n=6, 10: number analyzed (Participants) | 6 | 10
  Triglycerides; Week 24; n=6, 10 | 0.547 (0.9273) | -0.458 (1.2066)
  Triglycerides; Week 48; n=3, 7: number analyzed (Participants) | 3 | 7
  Triglycerides; Week 48; n=3, 7 | 0.260 (0.3894) | -0.486 (1.3993)
  Triglycerides; Week 60; n=2, 5: number analyzed (Participants) | 2 | 5
  Triglycerides; Week 60; n=2, 5 | 0.590 (0.8344) | -0.580 (1.0562)
  Triglycerides; Week 72; n=0, 1: number analyzed (Participants) | 0 | 1
  Triglycerides; Week 72; n=0, 1 |  | -0.240 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Urea/BUN; Baseline; n=14, 16 | 5.64 (1.167) | 5.72 (2.324)
  Urea/BUN; Day 8; n=13, 15: number analyzed (Participants) | 13 | 15
  Urea/BUN; Day 8; n=13, 15 | 0.04 (1.233) | -0.43 (1.252)
  Urea/BUN; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Urea/BUN; Day 28; n=13, 16 | -0.23 (1.678) | -0.13 (1.875)
  Urea/BUN; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Urea/BUN; Week 8; n=11, 16 | -0.09 (1.200) | -0.59 (1.985)
  Urea/BUN; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Urea/BUN; Week 12; n=12, 14 | 0.25 (1.270) | -0.50 (1.676)
  Urea/BUN; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Urea/BUN; Week 16; n=10, 16 | -0.05 (1.787) | -1.00 (1.304)
  Urea/BUN; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Urea/BUN; Week 24; n=11, 15 | -0.09 (1.200) | -0.27 (1.841)
  Urea/BUN; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Urea/BUN; Week 32; n=11, 14 | -0.55 (1.150) | 0.57 (1.708)
  Urea/BUN; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Urea/BUN; Week 40; n=8, 12 | -0.19 (1.387) | 0.29 (1.339)
  Urea/BUN; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Urea/BUN; Week 48; n=8, 13 | 0.38 (1.157) | 0.88 (1.927)
  Urea/BUN; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Urea/BUN; Week 60; n=5, 12 | 0.30 (0.908) | 0.54 (1.888)
  Urea/BUN; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Urea/BUN; Week 72; n=3, 4 | 0.50 (0.500) | 0.50 (0.408)
  Urea/BUN; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Urea/BUN; Week 84; n=0, 1 |  | 0.00 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

27. Secondary Outcome: Change From Baseline in Creatinine Clearance
Description: Creatinine clearance was calculated using Cockcroft-Gault formula. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline, Day 8, Day 28, Week 8, Week 16, Week 24, Week 32 and Week 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Milliliters per minute
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Milliliters per minute
  Baseline; n=14, 16 | 106.8 (31.79) | 104.8 (36.96)
  Day 8; n=1, 0: number analyzed (Participants) | 1 | 0
  Day 8; n=1, 0 | -13.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant. |
  Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28; n=13, 16 | -10.5 (13.06) | -10.4 (13.06)
  Week 8; n=0, 1: number analyzed (Participants) | 0 | 1
  Week 8; n=0, 1 |  | -12.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Week 16; n=10, 15: number analyzed (Participants) | 10 | 15
  Week 16; n=10, 15 | -7.3 (12.00) | -12.5 (16.41)
  Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24; n=11, 15 | -2.3 (13.94) | -13.9 (17.38)
  Week 32; n=9, 14: number analyzed (Participants) | 9 | 14
  Week 32; n=9, 14 | -1.4 (8.82) | -16.0 (16.31)
  Week 48; n=6, 12: number analyzed (Participants) | 6 | 12
  Week 48; n=6, 12 | -6.8 (17.61) | -16.5 (14.34)

28. Secondary Outcome: Change From Baseline in Lipase Levels
Description: Blood samples were collected for the analysis of clinical chemistry parameters such as lipase level. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Units per liter
  Lipase; Baseline; n=14, 16 | 29.1 (12.37) | 34.0 (18.54)
  Lipase; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Lipase; Day 8; n=14, 15 | 3.4 (9.19) | 12.5 (32.97)
  Lipase; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Lipase; Day 28; n=13, 16 | 3.3 (9.18) | 17.7 (63.64)
  Lipase; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Lipase; Week 8; n=11, 16 | 2.6 (8.65) | 13.6 (42.89)
  Lipase; Week 12; n=11, 14: number analyzed (Participants) | 11 | 14
  Lipase; Week 12; n=11, 14 | -2.4 (8.91) | 3.0 (19.24)
  Lipase; Week 16; n=10, 16: number analyzed (Participants) | 10 | 16
  Lipase; Week 16; n=10, 16 | 7.6 (13.94) | -0.8 (12.90)
  Lipase; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Lipase; Week 24; n=11, 15 | -2.7 (9.91) | 10.5 (29.18)
  Lipase; Week 32; n=11, 14: number analyzed (Participants) | 11 | 14
  Lipase; Week 32; n=11, 14 | 0.8 (9.82) | 20.6 (49.70)
  Lipase; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Lipase; Week 40; n=8, 12 | 0.6 (8.53) | 5.6 (19.78)
  Lipase; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Lipase; Week 48; n=8, 13 | 3.8 (6.18) | 3.4 (16.05)
  Lipase; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Lipase; Week 60; n=5, 12 | 5.0 (8.40) | 5.9 (22.01)
  Lipase; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Lipase; Week 72; n=3, 4 | 16.0 (14.11) | 41.0 (94.20)
  Lipase; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Lipase; Week 84; n=0, 1 |  | -9.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

29. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet and White Blood Cell (WBC) Count
Description: Blood samples were collected for the analysis of hematology parameters such as basophils, eosinophils. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Giga cells per liter
  Basophils; Baseline; n=14, 16 | 0.016 (0.0122) | 0.015 (0.0126)
  Basophils; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Basophils; Day 8; n=14, 15 | 0.006 (0.0134) | 0.002 (0.0094)
  Basophils; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Basophils; Day 28; n=13, 16 | 0.005 (0.0176) | 0.004 (0.0222)
  Basophils; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Basophils; Week 8; n=11, 16 | -0.001 (0.0122) | 0.004 (0.0120)
  Basophils; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Basophils; Week 12; n=12, 14 | -0.001 (0.0144) | 0.000 (0.0124)
  Basophils; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Basophils; Week 16; n=12, 16 | -0.002 (0.0147) | 0.005 (0.0137)
  Basophils; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Basophils; Week 24; n=11, 15 | 0.001 (0.0158) | 0.007 (0.0188)
  Basophils; Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Basophils; Week 32; n=11, 13 | 0.002 (0.0108) | 0.005 (0.0185)
  Basophils; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Basophils; Week 40; n=8, 12 | -0.000 (0.0207) | 0.003 (0.0144)
  Basophils; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Basophils; Week 48; n=8, 13 | 0.006 (0.0130) | 0.008 (0.0174)
  Basophils; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Basophils; Week 60; n=5, 12 | -0.002 (0.0164) | 0.004 (0.0173)
  Basophils; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Basophils; Week 72; n=3, 4 | -0.003 (0.0153) | 0.008 (0.0275)
  Basophils; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Basophils; Week 84; n=0, 1 |  | 0.010 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Eosinophils; Baseline; n=14, 16 | 0.087 (0.0935) | 0.158 (0.1681)
  Eosinophils; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Eosinophils; Day 8; n=14, 15 | 0.016 (0.0388) | 0.005 (0.1076)
  Eosinophils; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Eosinophils; Day 28; n=13, 16 | 0.023 (0.0253) | 0.033 (0.1939)
  Eosinophils; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Eosinophils; Week 8; n=11, 16 | 0.041 (0.0561) | 0.090 (0.1464)
  Eosinophils; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Eosinophils; Week 12; n=12, 14 | 0.023 (0.0492) | 0.240 (0.4390)
  Eosinophils; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Eosinophils; Week 16; n=12, 16 | 0.024 (0.0887) | 0.141 (0.3009)
  Eosinophils; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Eosinophils; Week 24; n=11, 15 | -0.003 (0.0987) | 0.159 (0.3737)
  Eosinophils; Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Eosinophils; Week 32; n=11, 13 | 0.016 (0.1108) | 0.075 (0.1921)
  Eosinophils; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Eosinophils; Week 40; n=8, 12 | -0.015 (0.1285) | 0.011 (0.1054)
  Eosinophils; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Eosinophils; Week 48; n=8, 13 | -0.028 (0.1241) | 0.122 (0.2186)
  Eosinophils; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Eosinophils; Week 60; n=5, 12 | -0.038 (0.1392) | 0.098 (0.2143)
  Eosinophils; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Eosinophils; Week 72; n=3, 4 | -0.043 (0.1185) | 0.053 (0.0660)
  Eosinophils; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Eosinophils; Week 84; n=0, 1 |  | 0.240 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Lymphocytes; Baseline; n=14, 16 | 1.656 (0.9039) | 1.418 (0.7921)
  Lymphocytes; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Lymphocytes; Day 8; n=14, 15 | 0.165 (0.4910) | 0.040 (0.3262)
  Lymphocytes; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Lymphocytes; Day 28; n=13, 16 | 0.132 (0.4841) | 0.297 (0.3042)
  Lymphocytes; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Lymphocytes; Week 8; n=11, 16 | 0.490 (0.5591) | 0.536 (0.6238)
  Lymphocytes; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Lymphocytes; Week 12; n=12, 14 | 0.417 (0.9401) | 0.525 (0.4922)
  Lymphocytes; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Lymphocytes; Week 16; n=12, 16 | 0.554 (0.6402) | 0.594 (0.7014)
  Lymphocytes; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Lymphocytes; Week 24; n=11, 15 | 0.271 (0.7466) | 0.647 (0.8692)
  Lymphocytes; Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Lymphocytes; Week 32; n=11, 13 | 0.173 (0.7166) | 0.818 (0.6910)
  Lymphocytes; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Lymphocytes; Week 40; n=8, 12 | 0.169 (0.6600) | 0.519 (0.6709)
  Lymphocytes; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Lymphocytes; Week 48; n=8, 13 | 0.474 (0.4207) | 0.563 (0.5703)
  Lymphocytes; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Lymphocytes; Week 60; n=5, 12 | 0.526 (0.3578) | 0.663 (0.6135)
  Lymphocytes; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Lymphocytes; Week 72; n=3, 4 | 0.673 (0.5327) | 0.623 (0.4280)
  Lymphocytes; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Lymphocytes; Week 84; n=0, 1 |  | 0.640 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Monocytes; Baseline; n=14, 16 | 0.367 (0.2075) | 0.306 (0.1117)
  Monocytes; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Monocytes; Day 8; n=14, 15 | 0.003 (0.2379) | 0.027 (0.1460)
  Monocytes; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Monocytes; Day 28; n=13, 16 | -0.042 (0.1999) | 0.031 (0.1196)
  Monocytes; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Monocytes; Week 8; n=11, 16 | -0.022 (0.1256) | 0.037 (0.1111)
  Monocytes; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Monocytes; Week 12; n=12, 14 | -0.053 (0.1215) | 0.065 (0.1075)
  Monocytes; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Monocytes; Week 16; n=12, 16 | -0.027 (0.1262) | 0.089 (0.1430)
  Monocytes; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Monocytes; Week 24; n=11, 15 | -0.067 (0.1152) | 0.017 (0.1716)
  Monocytes; Week 32; n=11, 13: number analyzed (Participants) | 11 | 14
  Monocytes; Week 32; n=11, 13 | -0.059 (0.1208) | 0.017 (0.1616)
  Monocytes; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Monocytes; Week 40; n=8, 12 | -0.030 (0.0685) | 0.011 (0.0983)
  Monocytes; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Monocytes; Week 48; n=8, 13 | -0.050 (0.1598) | 0.018 (0.0985)
  Monocytes; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Monocytes; Week 60; n=5, 12 | -0.088 (0.1359) | -0.003 (0.1305)
  Monocytes; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Monocytes; Week 72; n=3, 4 | 0.003 (0.0987) | 0.055 (0.1196)
  Monocytes; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Monocytes; Week 84; n=0, 1 |  | -0.230 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Total neutrophils; Baseline; n=14, 16 | 2.327 (1.2068) | 1.869 (1.0565)
  Total neutrophils; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Total neutrophils; Day 8; n=14, 15 | 0.090 (0.9029) | 0.072 (0.6338)
  Total neutrophils; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Total neutrophils; Day 28; n=13, 16 | 0.196 (0.7017) | 0.659 (0.9376)
  Total neutrophils; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Total neutrophils; Week 8; n=11, 16 | 0.480 (0.7919) | 0.344 (0.7325)
  Total neutrophils; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Total neutrophils; Week 12; n=12, 14 | 0.022 (0.5946) | 0.357 (0.5410)
  Total neutrophils; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Total neutrophils; Week 16; n=12, 16 | 0.780 (1.7187) | 1.030 (0.7759)
  Total neutrophils; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Total neutrophils; Week 24; n=11, 15 | -0.128 (0.7851) | 0.746 (1.3053)
  Total neutrophils; Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Total neutrophils; Week 32; n=11, 13 | 0.213 (0.9525) | 0.875 (1.0945)
  Total neutrophils; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Total neutrophils; Week 40; n=8, 12 | 0.224 (1.0274) | 0.390 (0.4501)
  Total neutrophils; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Total neutrophils; Week 48; n=8, 13 | 0.144 (0.5807) | 0.986 (1.0983)
  Total neutrophils; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Total neutrophils; Week 60; n=5, 12 | 0.162 (0.7959) | 1.507 (1.7191)
  Total neutrophils; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Total neutrophils; Week 72; n=3, 4 | 0.783 (1.6101) | 2.363 (2.0072)
  Total neutrophils; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Total neutrophils; Week 84; n=0, 1 |  | 2.060 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  Platelet; Baseline; n=14, 16 | 173.0 (65.30) | 176.9 (56.97)
  Platelet; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Platelet; Day 8; n=14, 15 | 21.6 (29.23) | 16.5 (29.08)
  Platelet; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Platelet; Day 28; n=13, 16 | 33.9 (29.87) | 30.8 (43.76)
  Platelet; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Platelet; Week 8; n=11, 16 | 57.8 (70.86) | 29.1 (57.51)
  Platelet; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Platelet; Week 12; n=12, 14 | 36.5 (33.68) | 39.2 (56.51)
  Platelet; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Platelet; Week 16; n=12, 16 | 35.7 (39.58) | 52.6 (56.43)
  Platelet; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Platelet; Week 24; n=11, 15 | 33.5 (31.41) | 58.7 (64.10)
  Platelet; Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Platelet; Week 32; n=11, 13 | 12.1 (33.87) | 55.6 (74.60)
  Platelet; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Platelet; Week 40; n=8, 12 | 25.6 (38.38) | 44.9 (48.17)
  Platelet; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Platelet; Week 48; n=8, 13 | 24.6 (36.49) | 53.5 (63.73)
  Platelet; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Platelet; Week 60; n=5, 12 | 43.0 (18.36) | 51.5 (58.12)
  Platelet; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Platelet; Week 72; n=3, 4 | 34.3 (40.15) | 64.0 (94.89)
  Platelet; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Platelet; Week 84; n=0, 1 |  | 88.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.
  WBC; Baseline; n=14, 16 | 4.44 (1.752) | 3.78 (1.522)
  WBC; Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  WBC; Day 8; n=14, 15 | 0.29 (1.082) | 0.15 (0.890)
  WBC; Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  WBC; Day 28; n=13, 16 | 0.33 (0.946) | 1.03 (1.105)
  WBC; Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  WBC; Week 8; n=11, 16 | 1.00 (1.015) | 1.02 (1.008)
  WBC; Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  WBC; Week 12; n=12, 14 | 0.42 (1.192) | 1.19 (1.005)
  WBC; Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  WBC; Week 16; n=12, 16 | 1.36 (2.050) | 1.86 (1.398)
  WBC; Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  WBC; Week 24; n=11, 15 | 0.09 (1.276) | 1.59 (2.075)
  WBC; Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  WBC; Week 32; n=11, 13 | 0.35 (1.264) | 1.78 (1.600)
  WBC; Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  WBC; Week 40; n=8, 12 | 0.36 (1.162) | 0.93 (0.965)
  WBC; Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  WBC; Week 48; n=8, 13 | 0.56 (0.655) | 1.70 (1.480)
  WBC; Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  WBC; Week 60; n=5, 12 | 0.58 (0.973) | 2.25 (1.579)
  WBC; Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  WBC; Week 72; n=3, 4 | 1.43 (1.210) | 3.10 (2.349)
  WBC; Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  WBC; Week 84; n=0, 1 |  | 2.70 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

30. Secondary Outcome: Change From Baseline in Hemoglobin Level
Description: Blood samples were collected for the analysis of hematology parameters such as hemoglobin. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Grams per liter
  Baseline; n=14, 16 | 132.9 (16.16) | 129.9 (21.08)
  Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Day 8; n=14, 15 | -1.0 (6.98) | -1.3 (4.37)
  Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28; n=13, 16 | -2.5 (8.76) | -0.9 (9.62)
  Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8; n=11, 16 | -4.5 (13.71) | 2.6 (12.48)
  Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12; n=12, 14 | -1.0 (12.59) | 2.1 (11.02)
  Week 16; n=12 16: number analyzed (Participants) | 12 | 16
  Week 16; n=12 16 | 0.0 (15.47) | 1.9 (10.14)
  Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24; n=11, 15 | -0.6 (10.60) | 1.5 (8.82)
  Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Week 32; n=11, 13 | -2.4 (10.66) | 1.5 (9.49)
  Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Week 40; n=8, 12 | -0.9 (12.14) | 0.7 (11.32)
  Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48; n=8, 13 | 0.0 (9.80) | 0.5 (13.48)
  Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60; n=5, 12 | -1.8 (13.99) | 5.0 (13.22)
  Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72; n=3, 4 | -4.3 (7.37) | 7.0 (8.72)
  Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84; n=0, 1 |  | -6.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

31. Secondary Outcome: Change From Baseline in Hematocrit Level
Description: Blood samples were collected for the analysis of hematology parameters such as hematocrit level. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Proportion of red blood cells in blood
  Baseline; n=14, 16 | 0.4024 (0.05259) | 0.3974 (0.06496)
  Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Day 8; n=14, 15 | -0.0015 (0.02666) | -0.0049 (0.01515)
  Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28; n=13, 16 | -0.0066 (0.03105) | -0.0043 (0.03313)
  Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8; n=11, 16 | -0.0105 (0.04383) | 0.0092 (0.04092)
  Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12; n=12, 14 | -0.0027 (0.03702) | 0.0054 (0.03419)
  Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16; n=12, 16 | -0.0033 (0.04275) | 0.0021 (0.03054)
  Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24; n=11, 15 | -0.0025 (0.03707) | 0.0062 (0.02787)
  Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Week 32; n=11, 13 | -0.0081 (0.03310) | 0.0062 (0.03144)
  Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Week 40; n=8, 12 | -0.0005 (0.03257) | 0.0063 (0.03601)
  Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48; n=8, 13 | 0.0065 (0.02919) | 0.0078 (0.04331)
  Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60; n=5, 12 | -0.0024 (0.04000) | 0.0200 (0.04520)
  Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72; n=3, 4 | -0.0170 (0.03119) | 0.0248 (0.02943)
  Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84; n=0, 1 |  | -0.0090 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

32. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume
Description: Blood samples were collected for the analysis of hematology parameters such as mean corpuscle volume. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Femtoliter
  Baseline; n=14, 16 | 99.1 (8.83) | 97.8 (9.28)
  Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Day 8; n=14, 15 | 0.1 (2.35) | 0.3 (1.71)
  Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28; n=13, 16 | 1.2 (3.26) | 0.3 (3.82)
  Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8; n=11, 16 | 0.3 (3.77) | -0.3 (6.02)
  Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12; n=12, 14 | 1.1 (7.73) | -1.5 (7.39)
  Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16; n=12, 16 | 0.3 (7.84) | -2.2 (8.85)
  Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24; n=11, 15 | -0.3 (8.25) | -2.0 (10.36)
  Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Week 32; n=11, 13 | -1.0 (8.54) | -2.4 (10.87)
  Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Week 40; n=8, 12 | 2.5 (8.75) | -0.7 (11.41)
  Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48; n=8, 13 | 2.0 (7.76) | -1.0 (11.73)
  Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60; n=5, 12 | 1.4 (7.89) | -1.2 (11.82)
  Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72; n=3, 4 | 0.3 (10.12) | 2.3 (14.10)
  Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84; n=0, 1 |  | 18.0 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

33. Secondary Outcome: Change From Baseline in Red Blood Cell Count
Description: Blood samples were collected for the analysis of hematology parameters such as RBC. Baseline was defined as the last pre-treatment value. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. NA indicates data was not available.
Time Frame: Baseline, Day 8, Day 28, Weeks 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | DTG 50 mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
Number analyzed (Participants) | 14 | 16
Trillion cells per liter
  Baseline; n=14, 16 | 4.09 (0.550) | 4.09 (0.731)
  Day 8; n=14, 15: number analyzed (Participants) | 14 | 15
  Day 8; n=14, 15 | 0.00 (0.254) | -0.04 (0.140)
  Day 28; n=13, 16: number analyzed (Participants) | 13 | 16
  Day 28; n=13, 16 | -0.08 (0.309) | -0.06 (0.318)
  Week 8; n=11, 16: number analyzed (Participants) | 11 | 16
  Week 8; n=11, 16 | -0.14 (0.434) | 0.12 (0.435)
  Week 12; n=12, 14: number analyzed (Participants) | 12 | 14
  Week 12; n=12, 14 | -0.05 (0.493) | 0.15 (0.477)
  Week 16; n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16; n=12, 16 | -0.03 (0.529) | 0.13 (0.478)
  Week 24; n=11, 15: number analyzed (Participants) | 11 | 15
  Week 24; n=11, 15 | 0.02 (0.464) | 0.18 (0.514)
  Week 32; n=11, 13: number analyzed (Participants) | 11 | 13
  Week 32; n=11, 13 | -0.04 (0.467) | 0.18 (0.504)
  Week 40; n=8, 12: number analyzed (Participants) | 8 | 12
  Week 40; n=8, 12 | -0.08 (0.392) | 0.09 (0.658)
  Week 48; n=8, 13: number analyzed (Participants) | 8 | 13
  Week 48; n=8, 13 | -0.00 (0.334) | 0.15 (0.625)
  Week 60; n=5, 12: number analyzed (Participants) | 5 | 12
  Week 60; n=5, 12 | -0.06 (0.428) | 0.28 (0.625)
  Week 72; n=3, 4: number analyzed (Participants) | 3 | 4
  Week 72; n=3, 4 | -0.20 (0.173) | 0.25 (0.759)
  Week 84; n=0, 1: number analyzed (Participants) | 0 | 1
  Week 84; n=0, 1 |  | -0.60 (NA) — Only one participant was analyzed for this treatment arm at this time point; thus, no standard deviation could be calculated for this single participant.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected in the time period from the first dose of study medication until early withdrawal or through the Week 48 analysis data cut-off date (median of 55 study weeks).
Description: SAEs and AEs were collected in members of Safety Population, comprised of all randomized participants who received at least one dose of study medication.
Groups:
- DTG 50mg BID: Participants received dolutegravir (DTG) 50 milligrams (mg) twice daily (BID) and the components of their current failing antiretroviral regimen, except raltegravir or elvitegravir, for 7 days during the Double-blind (DB) Phase. From Day 8, all participants continued to receive DTG 50 mg BID with an optimized background regimen in the Open-label Phase.
Arm/Group | DTG 50mg BID | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase
All-Cause Mortality (participants affected / at risk) | 2/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/14 | 4/16
Other Adverse Events (participants affected / at risk) | 11/14 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50mg BID (N=14) | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase (N=16)
Coronary artery disease (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Cardiac death (General disorders) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50mg BID (N=14) | Placebo BID in DB Phase; DTG 50 mg BID in Open-label Phase (N=16)
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 3
Dry eye (Eye disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Injection site induration (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal abscess (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Amnesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Ejaculation delayed (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.